CLINICAL TRIAL: NCT05626348
Title: The Clinical Study to Observe the Efficacy and Safety of Immunomodulators in Rheumatoid Arthritis Patients for 6 Months Treatment in China
Brief Title: The Clinical Efficacy of Immunomodulators in RA Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Qiang Shu, Chief Physician, Qilu Hospital of Shandong University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Response of DMARDs in RA QiluH
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Arthritis, Rheumatoid
Keywords: csDMARDs; TNFi
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — iguratimod; glucose utilization inhibitor; T 614; Methotrexate; Adalimumab; Leflunomide; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Methotrexate(MTX)+Iguratimod(IGU) (Experimental): Drug: Iguratimod（IGU），25mg, po, twice per day (Bid) prescribed at the beginning and adjusted due to patient response.
  Drug: Methotrexate(MTX)，10mg, po, quaque week (qw) prescribed at the beginning and adjusted due to patient response.
  For RA patients with naive or csDMARDs-IR
  Interventions: Drug: Iguratimod; Drug: Methotrexate
- Adalimumab+Methotrexate(MTX) (Experimental): Drug: Adalimumab，40mg, iH,q2w, once two weeks (q2w) prescribed at the beginning and adjusted due to patient response.
  Drug: Methotrexate(MTX)，7-10mg, po, quaque week (qw) prescribed at the beginning and adjusted due to patient response.
  For RA patients with csDMARDs-IR
  Interventions: Drug: Methotrexate; Drug: Adalimumab Injection
- Iguratimod(IGU)+Leflunomide(LEF)+Hydroxychloroquine(HCQ) (Experimental): Drug: Iguratimod（IGU），25mg, po, twice per day (Bid) prescribed at the beginning and adjusted due to patient response.
  Drug: Leflunomide(LEF)，20mg, po, quaque day (qd) prescribed at the beginning and adjusted due to patient response.
  Drug: Hydroxychloroquine(HCQ)，200mg, po, twice per day (Bid) prescribed at the beginning and adjusted due to patient response.
  For RA patients with csDMARDs-IR
  Interventions: Drug: Iguratimod; Drug: Leflunomide; Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Iguratimod — Iguratimod tablet，25mg, po, twice per day (Bid) prescribed at the beginning and adjusted due to patient response. Then may titer down until the endpoint.
  Other Names: IGU; T-614
  Arms: Iguratimod(IGU)+Leflunomide(LEF)+Hydroxychloroquine(HCQ); Methotrexate(MTX)+Iguratimod(IGU)
Drug: Methotrexate — Methotrexate，10mg, po, quaque week (qw) prescribed at the beginning and adjusted due to patient response. Then may titer down until the endpoint.
  Other Names: MTX
  Arms: Adalimumab+Methotrexate(MTX); Methotrexate(MTX)+Iguratimod(IGU)
Drug: Adalimumab Injection — Adalimumab Injection，40mg，iH，every two weeks (q2w) prescribed at the beginning and adjusted due to patient response. Then may titer down until the endpoint.
  Other Names: adalimu
  Arms: Adalimumab+Methotrexate(MTX)
Drug: Leflunomide — Leflunomide，20mg, po, quaque day (qd) prescribed at the beginning and adjusted due to patient response. Then may titer down until the endpoint.
  Other Names: LEF
  Arms: Iguratimod(IGU)+Leflunomide(LEF)+Hydroxychloroquine(HCQ)
Drug: Hydroxychloroquine — Hydroxychloroquine，200mg, po, twice per day (bid) prescribed at the beginning and adjusted due to patient response. Then may titer down until the endpoint.
  Other Names: HCQ
  Arms: Iguratimod(IGU)+Leflunomide(LEF)+Hydroxychloroquine(HCQ)

SUMMARY:
This study includes naive patients and csDMARDs-IR RA patients, treated with different regimens such as Iguratimod combination of different csDMARDs, or csDMARD with TNF inhibitors for 24 weeks. The disease activity and drug response will be observed. The immune disorder and synovial function will be evaluated at the same time.

DETAILED DESCRIPTION:
In this study cohorts, naïve or csDMARDs-IR patients are treated with different csDMARDs combination or TNF inhibitors for 24 weeks to get remission in clinical. The biomarkers in their plasma and synovial fluid and tissue specimens from RA patients are screened to predict the efficacy of specific treatment.

ELIGIBILITY:
Inclusion Criteria:

-

1.Patients with RA who meet ACR 1987 rheumatoid arthritis classification criteria or ACR/EULAR 2010 rheumatoid arthritis Classification Criteria and have knee dysfunction.

1. ACR 1987 rheumatoid arthritis classification criteria

   1. morning stiffness lasting at least 1 hour (≥6w)
   2. there are 3 or more joint areas swollen (≥6w)
   3. swelling of the wrist, metacarpophalangeal, and proximal phalangeal joint areas (≥6w)
   4. symmetrical arthrogryposis (≥6w)
   5. hand x-ray changes (at least osteoporosis and joint space narrowing)
   6. positive rheumatoid factor (titer > 1:32) RA can be diagnosed by meeting 4 of the above 7 items
2. ACR/EULAR 2010 rheumatoid arthritis Classification Criteria

   1. Involved joints

      - 1 large joint (0 points)
      * 2-10 large joints (1 point)
      * 1-3 small joints (with or without large joints) (2 points)
      * 4-10 small joints (with or without large joints) (3 points)
      * more than 10 small joints (at least one small joint) (5 points)
   2. Serological indicators

      * RF and ACPA negative (0 points)
      * RF and ACPA, at least one of which is low titer positive. (2 points)
      * RF and ACPA with at least one high titer positive (3 points)
   3. Acute chronotropic reactants

      * Both CRP and ESR normal (0 points)
      * Abnormal CRP or ESR (1 point)
   4. Duration of synovitis

      * <6 weeks (0 points)
      * ≥6 weeks (1 point)

        2.Patients with OA who meet the 1995 Classification Criteria for OA and have knee dysfunction 1995 Classification Criteria for Osteoarthritis of the Knee Clinical criteria

        a. Knee pain most of the time in the last 1 month b. Bone rubbing sound c, morning stiffness ≤ 30 minutes d, age ≥ 38 years e, with bony enlargement Knee OA can be diagnosed if a+b+c+d or a+b+e is met

        3.Age-sex matched healthy volunteers who checked in our hospital.

        4.Age > 18 years old;

        5.Voluntarily participate in this study and sign an informed consent form

Exclusion Criteria:

1. Patients with combined active hepatitis
2. Patients with active tuberculosis
3. Patients withinfection and malignancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-12-22 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients who achieve clinical remission using European League Against Rheumatism (EULAR) response criteria DAS28. | week 24
  The percentage of patients whose Disease Activity Score in 28 Joints (DAS28) achieve remission（DAS28-ESR≤ 2.6）and Low Disease Activity (DAS28-ESR ≤ 3.2). The DAS28 is a composite score derived from 4 of these measures，that is the count of tender joint count（TJC, 0-28）and swollen joint count（SJC, 0-28）, measure erythrocyte sedimentation rate (ESR, mm/h) or C reactive protein (CRP, mg/L) and to make a patient assessment of disease activity i.e. 'global assessment of health' (GH) using a 100 mm visual analogue scale (VAS) with 0 = best, 100 = worst. DAS28 values were calculated as follows: DAS28- ESR = 0.56√(TJC) + 0.28√(SJC) + 0.70 ln ESR + 0.014 x GH. High disease activity: DAS28-ESR > 5.1; Moderate disease activity: 5.1≥ DAS28 > 3.2 to 5.1; Low disease activity (LDA) and Remission mean Clinical remission.

SECONDARY OUTCOMES:
The percentage of patients who achieve clinical remission using DAS28-ESR. | week 12
  The percentage of patients whose DAS28 achieve remission（DAS28-ESR≤ 2.6）and Low Disease Activity (DAS28-ESR ≤ 3.2) .
Percentage of Disease Activity Score 28 (DAS28) -ESR Criteria Responders | baseline,week 12,week 24
  △DAS28 indicates the decline of DAS28-ESR from the baseline to week 30. EULAR response states were classified as follows: good responders were patients with an improvement from baseline (△DAS28-ESR) of > 1.2 and a DAS28-ESR at week 30 ≤ 3.2. Moderate responders: △DAS28 > 1.2 and still DAS28 > 3.2 at week 30, or 1.2 ≥△DAS28 > 0.6 and DAS28 ≤ 5.1 at week 30. Nonresponders：△DAS28 ≤0.6 or DAS28 >5.1 at week 30. DAS28-defined remission was classified as a score of <2.6.
Percentage of participants achieving ACR/EULAR remission | week 12,week 24
  If all of the following 4 parameters are fulfilled, it is defined as remission: TJC ≤ 1, SJC ≤ 1, CRP ≤ 1 mg/dL, Patient global assessment（PGA） ≤ 1 cm (on a visual analog scale ranging from 0-10 cm, with higher scores indicating severe disease).
Change from baseline Simplified Disease Activity Index (SDAI) | up to week 24
  The SDAI is a composite score derived from these measures，that is the count of tender joint count（TJC, 0-28）, swollen joint count（SJC, 0-28）, C-reactive protein (CRP, mg/L), Patient global assessment（PGA）and physician global assessment（PHGA）, each of the last two was assessed on a visual analog scale ranging from 0-10 cm, with higher scores indicating severe disease. SDAI score will be calculated with formula SDAI = TJC + SJC + PGA+PHGA+ CRP. SDAI score exceeding 26 is considered high disease activity; 11 <SDAI ≤26，moderate disease activity; 3.3 <SDAI ≤11, low disease activity; remission is SDAI score ≤ 3.3.
Change from baseline Clinical Disease Activity Index (CDAI) | up to week 24
  Change from baseline Clinical Disease Activity Index (CDAI) CDAI is a composite score derived from these measures，that is the count of tender joint count（TJC, 0-28）, swollen joint count（SJC, 0-28）, Patient global assessment（PGA）and physician global assessment（PHGA）, each of the last two was CDAI score will be calculated with formula CDAI = TJC + SJC + PGA + PHGA. CDAI > 22 is considered high disease activity; 10 <CDAI ≤ 22, moderate disease activity; 2.8 <CDAI ≤10, low disease activity; remission is CDAI score ≤2.8.
Change From Baseline in C-reactive Protein (CRP) | up to week 24
  Change from Baseline in C-reactive Protein (CRP), a component index of ACR20 and SDAI, CRP will be measured with blood samples.
Change From Baseline in Erythrocyte Sedimentation Rate (ESR) | up to week 24
  Change from Baseline in ESR, that is a component index of ACR20, DAS28-ESR and SDAI, ESR will be measured with blood samples.
Change from baseline Health Assessment Questionnaire Disability Index (HAQ-DI) | up to week 24
  hange from Baseline in HAQ-DI, a participant assessed measure of health assessment, shaveing eight dimensions of functional activity: pruning, dressing, rising, eating, walking, personal hygiene, reach, grip, and other routine activities. Each item on a single scale has 4 degrees ranging from 0 (no functional difficulty) to 3 (unable to do), with higher scores indicating severe disease.
Percentage of American College of Rheumatology [ACR] 20、 [ACR]50、 [ACR]70 Criteria Responders every time | up to week 24
  Percentage of American College of Rheumatology [ACR] 20、 [ACR]50、 [ACR]70 Criteria Responders every time.
Incidence of participant withdrawal | up to week 24
  Percentage of participants who withdraw from this study.
Number of participants with"adverse events (AEs)" | up to week 24
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Number of participants with"adverse events (AEs)"i.e. physical exam abnormalities，vital sign abnormalities，laboratory value abnormalities，symptom or disease (new or exacerbated) temporally associated with the use of a medicinal product.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyun Yang, Study Director — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Jinan, Shandong, China